CLINICAL TRIAL: NCT02892916
Title: The Prevention of Post Operative Cognitive Dysfunction by Ketamine: a Prospective Multicenter Randomized Blinded Placebo-controlled Trial in Elderly Patients Undergoing Elective Orthopaedic Surgery
Brief Title: Ketamine and Postoperative Cognitive Dysfunction
Acronym: POCK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P150910; 2016-000691-16 (EudraCT Number); PHRC-15-15-0534 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2016-07-31; First posted 2016-09-08 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Post Operative Cognitive Dysfunction
Keywords: Post-operative cognitive dysfunction (POCD); Delirium; Ketamine; Elective orthopaedic surgery
MeSH Terms: conditions — Delirium | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Patients in this experimental group will receive a bolus of low intravenous dose (sub-anaesthetic) 0.5 mg/kg ketamine following induction of anaesthesia.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Patients in this control group will receive a bolus of an intravenous normal saline solution following induction of anaesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — A bolus of low intravenous dose (sub-anaesthetic) 0.5 mg/kg ketamine following induction of anaesthesia.
  Other Names: Ketamine hydrochloride
  Arms: Ketamine
Drug: Placebo — A bolus of an intravenous normal saline solution following induction of anaesthesia.
  Other Names: Normal saline solution
  Arms: Placebo

SUMMARY:
Over 30 million patients require a major surgery annually in the US alone and more than half of them are performed in patients over 60 years of age. Post-operative cognitive dysfunction (POCD) is a keystone complication of these surgeries and affects up to 40% of surgical patients aged over 60 years on discharge from the hospital. Despite controlled longitudinal studies have shown that POCD is transient, it is associated with delirium, higher mortality, earlier retirement, and greater utilization of social financial assistance The pathophysiology of persistent postoperative cognitive dysfunction and causal relationship between POCD and delirium remain incompletely understood. Identified clinical risk factors for both include advanced age, type of surgery, preexisting cognitive impairment, and drug addiction. We and others have provided evidence that the inflammatory response triggered by surgical trauma and pain may contribute to the development of delirium and cognitive impairment after surgery.

Ketamine, a N-methyl-D-aspartic acid receptor antagonist, is commonly used in anaesthesia and postoperative analgesia. By reducing both pain and glutamate excitotoxic effects on neuronal and microglial brain cells, it contributes to tone down the neuroinflammatory process associated with surgery. A recent body of evidence has shown that ketamine reduces the depressive-like behavior induced by inflammatory or stress-induced stimuli in mice. Ketamine was also found to reduce levels of inflammatory biomarkers in cardiac surgical patients.

Orthopaedic surgery is a high-risk situation for developing postoperative cognitive dysfunction. In patients undergoing non-cardiac surgery, the prevalence of POCD is 26% one week after surgery and decreased to 10% at 3 months postoperatively, and a similar prevalence is found 12 months after the operation. Postoperative delirium is associated with an increased risk of POCD. Hundred thousands of patients > 60 years undergo elective orthopaedic procedures per year around the world.

DETAILED DESCRIPTION:
The design consists in a prospective multicenter randomized blinded placebo-controlled trial in elderly patients undergoing elective orthopaedic surgery.

Patients will be informed at the pre-anaesthetic consultation, 7 to 30 days before surgery. They will be randomized the day before surgery. Cognitive and depressive status at baseline will be assessed precisely the day pior to surgery with cognitive tests. Self-administered scores will be recorded to evaluate depression, anxiety, and quality of life.

At the day of surgery, patients in the experimental group will receive a bolus of low intravenous dose (sub-anaesthetic) 0.5 mg/kg ketamine following induction of anaesthesia. Patients in the control group will receive a bolus of an intravenous normal saline solution following induction of anaesthesia.

From D0 (2 hours after surgery end) to D7 or discharge from the hospital if earlier, delirium, pain, adverse clinical and psychiatric events will be measured and recorded.

Cognitive functions, neuropathic pain, depression, anxiety and quality of life will be assessed at D7 or discharge from the hospital if earlier and D90.

Inflammatory markers will be measured before surgery, at D1, D7 or discharge from the hospital if earlier and D90.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 60 years and older
2. Competent to provide informed consent
3. Undergoing major elective orthopaedic surgery under general anaesthesia
4. Patients with and without pre-existing neurodegenerative disease

Exclusion Criteria:

1. Moribund patient or patient under palliative care
2. Expected length of stay at hospital < 48 hours
3. Patient under tutorship or curatorship
4. Surgical procedure performed under spinal or epidural anaesthesia without general anaesthesia
5. Emergency surgery (i.e. emergency hip fracture)
6. Patients with a known allergy to ketamine
7. Contraindication for ketamine: severe, uncontrolled arterial hypertension or severe heart (FEVG<25%)
8. Patient with glaucoma or history of thyrotoxicosis
9. Severe audition or vision disorder
10. Patients with drug misuse history (e.g., ketamine, cocaine, heroin, amphetamine, methamphetamine, MDMA (methylenedioxymethamphetamine), phencyclidine, lysergic acid, mescaline, psilocybin)
11. Patients taking anti-psychotic medications (e.g., chlorpromazine, clozapine, olanzapine, risperidone, haloperidol, quetiapine, risperidone, paliperidone, amisulpride, sertindole)
12. Patients with severe alcohol liver disease (TP<50% and or bilirubin > 50 µmol/L)
13. Pregnant or breast-feeding woman
14. Patient not speaking French
15. Absence of informed consent or request to not participate to the study
16. Non affiliation to the social security

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of early postoperative cognitive dysfunction | Days 7 and 90 after surgery
  POCD assessed using MoCA (Montreal Cognitive Assessment) test and others cognitive tests included in the calculation of the combined Z-score

SECONDARY OUTCOMES:
Post-operative cognitive dysfunction type | Days 7 and 90 after surgery
  The evaluation should be based on differences between pre- and postoperative performance (7 days or at discharge from the hospital if earlier and 3 months or earlier at the surgical follow-up visit depending on the practices of the different centers).
Post-operative cognitive dysfunction severity | Days 7 and 90 after surgery
  The evaluation should be based on differences between pre- and postoperative performance (7 days or at discharge from the hospital if earlier and 3 months or earlier at the surgical follow-up visit depending on the practices of the different centers).
The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) | Days 7 before surgery or discharge from the hospital
  Measurements will start from postoperative day 0 two hours after the end of surgery to day 7 or discharge from the hospital if earlier, twice daily (morning and evening) with at least 6 hours between two consecutive measurements.
Early postoperative delirium | 7 days after surgery
  Patients with at least one episode of delirium measured by CAM (Confusion Assessment Method) or CAM-ICU (adaptation used in Intensive Care Unit) scores between day 0 and day 7
Depression | Days 7 and 90 after surgery
  Depression assessed using the Geriatric Depression Scale (GDS)
Anxiety | Days 7 and 90 after surgery
  Anxiety assessed using the Hospital and Anxiety Depression Scale.
Pain status: Visual Analog Scale | Day prior to surgery, at days 7 and 90 after surgery
  Pain scores assessed by the patient-reported Visual Analog Scale. Neuropathic pain at 3 months measured by the DN4 (Douleur Neuropathique en 4 questions) questionnaire.
Time from surgery to POCD. | Days 7 and 90 after surgery
  Time of occurrence of POCD (early or late) and his association with postoperative delirium
Pre-existing cognitive status | Days 7 and 90 after surgery
  Pre-existing cognitive status measured by the preoperative combined Z-score for cognitive functions and his association with the occurrence of postoperative delirium
Preoperative Charlson's score for comorbidities | Days 7 and 90 after surgery
  Preoperative Charlson's sore for comorbidities and his association with the occurrence of postoperative delirium
Intraoperative serious adverse events | Day 7
  Intraoperative serious adverse events such as bleeding requiring at least 2 red cell units or unexpected prolonged duration of surgery and their association with postoperative delirium.
Postoperative adverse events | Day 7
  Early post-operative complications (reoperation, hospital readmission, bleeding, transfusion, sepsis, hypoxemia, sodium disorders, specific medications, presence or absence of a specific rehabilitation program) recorded from patients' charts and their association with postoperative delirium.
Hospital length of stay | Day 90
  Hospital length of stay assessed from patients' medical administrative data in days
Cause of death | Day 90
  Cause of death as postoperative cardio-respiratory arrest and degradation of the general condition
Hospital readmission | Day 90
  Hospital readmission during the follow up, whatever the etiology
Inflammatory biomarkers | Day 90
  Inflammatory biomarkers (C Reactive Protein, Interleukin-6, Interleukin-2, TNFalpha, B-type natriuretic peptide and Troponin) levels and their association with the occurrence of postoperative delirium and long term POCD
Quality of life evaluated thanks to the SF-36 scale | Day 90
  Quality of life evaluated thanks to the SF-36 scale is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state

CONTACTS AND LOCATIONS:
Overall Officials: Franck Verdonk, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP - Hôpital Saint-Antoine, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurdi MS, Theerth KA, Deva RS. Ketamine: Current applications in anesthesia, pain, and critical care. Anesth Essays Res. 2014 Sep-Dec;8(3):283-90. doi: 10.4103/0259-1162.143110. PMID 25886322
- [Background] Jabre P, Combes X, Lapostolle F, Dhaouadi M, Ricard-Hibon A, Vivien B, Bertrand L, Beltramini A, Gamand P, Albizzati S, Perdrizet D, Lebail G, Chollet-Xemard C, Maxime V, Brun-Buisson C, Lefrant JY, Bollaert PE, Megarbane B, Ricard JD, Anguel N, Vicaut E, Adnet F; KETASED Collaborative Study Group. Etomidate versus ketamine for rapid sequence intubation in acutely ill patients: a multicentre randomised controlled trial. Lancet. 2009 Jul 25;374(9686):293-300. doi: 10.1016/S0140-6736(09)60949-1. Epub 2009 Jul 1. PMID 19573904
- [Background] Riou B, Lecarpentier Y, Viars P. Inotropic effect of ketamine on rat cardiac papillary muscle. Anesthesiology. 1989 Jul;71(1):116-25. doi: 10.1097/00000542-198907000-00020. PMID 2751123
- [Background] Riou B, Viars P, Lecarpentier Y. Effects of ketamine on the cardiac papillary muscle of normal hamsters and those with cardiomyopathy. Anesthesiology. 1990 Nov;73(5):910-8. doi: 10.1097/00000542-199011000-00019. PMID 2240681
- [Background] Zanos P, Moaddel R, Morris PJ, Georgiou P, Fischell J, Elmer GI, Alkondon M, Yuan P, Pribut HJ, Singh NS, Dossou KS, Fang Y, Huang XP, Mayo CL, Wainer IW, Albuquerque EX, Thompson SM, Thomas CJ, Zarate CA Jr, Gould TD. NMDAR inhibition-independent antidepressant actions of ketamine metabolites. Nature. 2016 May 26;533(7604):481-6. doi: 10.1038/nature17998. Epub 2016 May 4. PMID 27144355
- [Background] Harraz MM, Tyagi R, Cortes P, Snyder SH. Antidepressant action of ketamine via mTOR is mediated by inhibition of nitrergic Rheb degradation. Mol Psychiatry. 2016 Mar;21(3):313-9. doi: 10.1038/mp.2015.211. Epub 2016 Jan 19. PMID 26782056
- [Background] Zorumski CF, Nagele P, Mennerick S, Conway CR. Treatment-Resistant Major Depression: Rationale for NMDA Receptors as Targets and Nitrous Oxide as Therapy. Front Psychiatry. 2015 Dec 9;6:172. doi: 10.3389/fpsyt.2015.00172. eCollection 2015. PMID 26696909
- [Background] Hudetz JA, Patterson KM, Iqbal Z, Gandhi SD, Byrne AJ, Hudetz AG, Warltier DC, Pagel PS. Ketamine attenuates delirium after cardiac surgery with cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2009 Oct;23(5):651-7. doi: 10.1053/j.jvca.2008.12.021. Epub 2009 Feb 23. PMID 19231245
- [Background] Arrowsmith JE, Harrison MJ, Newman SP, Stygall J, Timberlake N, Pugsley WB. Neuroprotection of the brain during cardiopulmonary bypass: a randomized trial of remacemide during coronary artery bypass in 171 patients. Stroke. 1998 Nov;29(11):2357-62. doi: 10.1161/01.str.29.11.2357. PMID 9804648
- [Derived] Verdonk F, Lambert P, Gakuba C, Nelson AC, Lescot T, Garnier F, Constantin JM, Saurel D, Lasocki S, Rineau E, Diemunsch P, Dreyfuss L, Tavernier B, Bezu L, Josserand J, Mebazaa A, Coroir M, Nouette-Gaulain K, Macouillard G, Glasman P, Lemesle D, Minville V, Cuvillon P, Gaudilliere B, Quesnel C, Abdel-Ahad P, Sharshar T, Molliex S, Gaillard R, Mantz J. Preoperative ketamine administration for prevention of postoperative neurocognitive disorders after major orthopedic surgery in elderly patients: A multicenter randomized blinded placebo-controlled trial. Anaesth Crit Care Pain Med. 2024 Aug;43(4):101387. doi: 10.1016/j.accpm.2024.101387. Epub 2024 May 6. PMID 38710325